CLINICAL TRIAL: NCT05839574
Title: Evaluation of the Therapeutic Effect of Adding Letrozole to the Protocol of Combined Treatment of Cesarean Scar Pregnancy
Brief Title: Letrozole add-on in the Treatment of Cesarean Scar Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Iwona Magdalena Gawron, M.D., Ph.D., Principal Investigator, Jagiellonian University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1072.6120.46.2021
Record Dates: First submitted 2023-04-15; First posted 2023-05-03 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Cesarean Scar Pregnancy
Keywords: cesarean scar pregnancy; operative hysteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTX in monotherapy (Active Comparator): Combined treatment with MTX followed by hysteroscopic evacuation of POC
  Interventions: Drug: MTX monotherapy
- MTX + letrozole add-on (Active Comparator): Combined treatment with MTX + letrozole add-on followed by hysteroscopic evacuation of POC
  Interventions: Drug: MTX + letrozole add-on

INTERVENTIONS:
Drug: MTX monotherapy — MTX in a single dose of 100 mg intravenously and 50 mg in intra-amniotic injection (day 0), along with 30 mg potassium chloride in case of positive fetal heartbeat (FH), and subsequent hysteroscopic evacuation of products of conception (POC)
  Arms: MTX in monotherapy
Drug: MTX + letrozole add-on — MTX in a single dose of 100 mg intravenously and 50 mg in intra-amniotic injection (day 0), along with 30 mg potassium chloride in case of positive fetal heartbeat (FH) + Letrozole in a daily dose of 5 mg (2 x 2.5 mg) orally for 10 days from day 0, and subsequent hysteroscopic evacuation of products of conception (POC)
  Arms: MTX + letrozole add-on

SUMMARY:
It is hypothesized that the inhibition of estradiol production by letrozole may interfere with physiological effects of progesterone necessary to maintain the pregnancy. There is no reference treatment of cesarean scar pregnancy (CSP) as the limited number of cases precludes the extrapolation of results. In our center we successfully use two-step treatment with methotrexate (MTX) followed by hysteroscopic removal of products of conception (POC). The time in between is needed to achieve a decrease in the trophoblast's vital potential (B-hCG fall) and its vascularization. Additional administration of letrozole could further reduce the vital potential of the pregnancy, eliminating the need for another dose of MTX, resulting in faster healing and lower rate of complications.

DETAILED DESCRIPTION:
A prospective cohort study is conducted among women with cesarean scar pregnancy (CSP). Women with increasing B-human chorionic gonadotropin (B-hCG) concentrations are included.

Two study arms were planned:

* women treated with a single dose of 100 mg MTX intravenously and 50 mg MTX in intra-amniotic injection (day 0), along with 30 mg potassium chloride in case of positive fetal heartbeat (FH)
* women treated with a single dose of 100 mg MTX intravenously and 50 mg MTX in intra-amniotic injection (day 0), along with 30 mg potassium chloride in case of positive fetal heartbeat (FH) with additional use of letrozole 5 mg orally (from day 0) for 10 days.

Blood parameters (B-hCG, hemoglobin, total blood count, creatinine, urea, alanine/aspartate transaminase, gamma-glutamyltransferase, bilirubin) were tested on days 0,4,7, followed by B-hCG concentration measurement every 7 days until surgery. After obtaining satisfactory decrease in B-hCG and POC vascularization, women underwent hysteroscopic evacuation of POC. Blood loss parameters, frequency of conversion from hysteroscopy to laparoscopy and laparotomy were measured.

The women were given the option to choose the treatment used in the study. All enrolled women gave informed written consent to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* CSP confirmed on pelvic ultrasound
* consent of the Bioethics Committee for termination of CSP
* increasing B-hCG concentrations

Exclusion Criteria:

* heterotopic pregnancy
* decreasing B-hCG concentrations

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Blood loss during the procedure expressed as a decrease in hemoglobin concentration | up to 6 months
  Decrease in hemoglobin concentration in g/dl on day 1 after the procedure compared to the pre-procedure concentration
Blood loss volume during the procedure expressed in volume units | up to 6 months
  The volume of blood lost during the procedure in ml
Conversion rate from hysteroscopy to laparoscopy or laparotomy due to due to hemorrhage | up to 6 months
  Percentage (%) of conversion from hysteroscopy to laparoscopy or laparotomy due to hemorrhage

SECONDARY OUTCOMES:
The effect of treatment on bone marrow function (red blood cells) | up to 6 months
  Change in red blood count (T/l) in the course of treatment (day 0,4,7)
The effect of treatment on bone marrow function (white blood cells) | up to 6 months
  Change in white blood count (G/l) in the course of treatment (day 0,4,7)
The effect of treatment on bone marrow function (platelets) | up to 6 months
  Change in platelet count (G/l) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (serum total bilirubin) | up to 6 months
  Changes in the concentrations of serum total bilirubin (mg/dl) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (alanine transaminase) | up to 6 months
  Changes in the concentrations of alanine transaminase (IU/l) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (aspartate transaminase) | up to 6 months
  Changes in the concentrations of aspartate transaminase (IU/l) in the course of treatment (day 0,4,7)
The effect of treatment on liver function (gamma-glutamyltransferase) | up to 6 months
  Changes in the concentrations of gamma-glutamyltransferase (IU/l) in the course of treatment (day 0,4,7)
The effect of treatment on kidneys function (urea) | up to 6 months
  Changes in the concentrations of serum urea (mmol/l) in the course of treatment (day 0,4,7)
The effect of treatment on kidneys function (creatinine) | up to 6 months
  Changes in the concentrations of serum and creatinine (mg/dl) in the course of treatment (day 0,4,7)

CONTACTS AND LOCATIONS:
Overall Officials: Iwona M. Gawron, M.D., Ph.D., Principal Investigator — Jagiellonian University; Robert Jach, Prof., Ph.D., Study Chair — Jagiellonian University
Locations (1):
- Jagiellonian University Medical College, Department of Gynecology and Obstetrics, Clinic of Gynecological Endocrinology, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No